CLINICAL TRIAL: NCT00175071
Title: Effect of Conventional and Reformulated Vegetable Oils for Use by the Snack Food Industry on Plasma Lipid Levels and Inflammatory Markers
Brief Title: Effect of Vegetable Oils for Use by the Snack Food Industry on Plasma Lipid Levels and Inflammatory Markers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tufts University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: HL54727-1537
Record Dates: First submitted 2005-09-08; First posted 2005-09-15 (Estimated); Last update posted 2018-07-13 (Actual); Status verified 2018-07

CONDITIONS: Hyperlipidemias; Metabolic Syndrome X; Cardiovascular Diseases
MeSH Terms: conditions — Hyperlipidemias; Metabolic Syndrome; Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- Comparison of cooking oils (Experimental): Postmenopausal women (50-85 y) with LDL cholesterol 120 mg/dL.
  Interventions: Behavioral: Comparison of cooking oils

INTERVENTIONS:
Behavioral: Comparison of cooking oils — 30 subjects will consume each of the two diets in randomized order for 5 weeks each. Diets will be designed to maintain body weight; will have 30% of energy as fat which 2/3 or 20% of energy will be either the conventional or reformulated fat. Blood lipids and C reactive protein (CRP) as well as indicators of how lipids are processed in the blood will be measured at the end of each dietary phase.

SUMMARY:
The current study is designed to assess the effect of a conventional cooking oil (hydrogenated oil) and a reformulated fat low in trans fatty acids on cardiovascular disease risk factors.

DETAILED DESCRIPTION:
It is known that in subjects with high cholesterol levels that substitution of hydrogenated fat (high in trans fat) with vegetable oil results in higher levels of total and LDL cholesterol ("bad" cholesterol). There has been tremendous interest within the food industry to identify cooking fats that have the physical properties necessary to make shelf stable products and have textural characteristics similar to existing products but that also favorably affects risk factors for coronary heart disease (CHD) such as LDL cholesterol levels and inflammatory markers. The current study is designed to assess the effect of a conventional cooking oil (hydrogenated oil) and a reformulated fat low in trans fatty acids on cardiovascular disease risk factors.

ELIGIBILITY:
Inclusion Criteria:

* Gender: female
* Age: 50-85 years
* LDL-C concentrations >120 mg/dL
* Menopausal status: postmenopausal

Exclusion Criteria:

* Use of medications known to affect lipid metabolism
* Untreated thyroid disease
* Diabetes mellitus
* Abnormal kidney function
* Abnormal liver function
* Smoking
* Alcohol consumption > 2 drinks/day

Ages: 50 Years to 85 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2004-03; Primary Completion 2007-04 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Serum lipid, lipoprotein and apolipoprotein concentrations, measures of inflammation, cholesteryl ester transfer protein (CETP) and lecithin-cholesterol acetyltransferase (LCAT) activities, endogenous lipid synthesis rates, expression of genes associated | 5 weeks period

CONTACTS AND LOCATIONS:
Overall Officials: Alice H Lichtenstein, D.Sc., Principal Investigator — Tufts Medical Center
Locations (1):
- Jean Mayer USDA Human Nutrition Research Center on Aging at Tufts University, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Vega-Lopez S, Matthan NR, Ausman LM, Ai M, Otokozawa S, Schaefer EJ, Lichtenstein AH. Substitution of vegetable oil for a partially-hydrogenated fat favorably alters cardiovascular disease risk factors in moderately hypercholesterolemic postmenopausal women. Atherosclerosis. 2009 Nov;207(1):208-12. doi: 10.1016/j.atherosclerosis.2009.03.039. Epub 2009 Apr 5. PMID 19423109
- See also: Click here for more information about this study: — http://hnrc.tufts.edu